CLINICAL TRIAL: NCT07011667
Title: Efficacy and Safety of Cagrilintide s.c. in Combination With Semaglutide s.c. (CagriSema s.c.) Once Weekly for Weight Management and Long-term Weight Maintenance in Participants With Obesity
Brief Title: A Research Study to Look at How Well CagriSema Helps People Living With Obesity Lose Weight and Maintain Weight Loss in the Long-term
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-8484; U1111-1318-6372 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-06-01; First posted 2025-06-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants in the main phase will be randomised in double blinded manner to receive either CagriSema or matching placebo. In the extension phase, eligible participants will be re-randomised and enter the open label extension phase. Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema (Experimental): Participants will receive CagriSema subcutaneously once weekly in a dose escalation manner (dose increases every 4 weeks) for up to 16 weeks followed by CagriSema maintenance dose subcutaneously once weekly for 64 weeks in the main phase of the study. Participants randomised to this arm will be included in the extension phase to receive 1 of the 3 dose levels of CagriSema for 80 weeks.
  Interventions: Drug: CagriSema (Cagrilintide B and Semaglutide I)
- Placebo (Placebo Comparator): Participants will receive placebo matched to CagriSema subcutaneously once weekly for 80 weeks in the main phase of the study. Participants randomised to this arm will be included in the extension phase to receive CagriSema with flexible dose escalation for 80 weeks.
  Interventions: Drug: CagriSema (Cagrilintide B and Semaglutide I); Drug: Placebo matched to CagriSema (Cagrilintide B and Semaglutide I)

INTERVENTIONS:
Drug: CagriSema (Cagrilintide B and Semaglutide I) — CagriSema (Cagrilintide B and Semaglutide I) will be administered subcutaneously using DV3384 pen-injector.
Drug: Placebo matched to CagriSema (Cagrilintide B and Semaglutide I) — Placebo matched to Cagrilintide B and placebo matched to Semaglutide I will be administered subcutaneously using DV3384 pen-injector.
  Arms: Placebo

SUMMARY:
This study will look at how well CagriSema helps people living with obesity to lose weight and maintain the weight loss long-term. The study has 2 parts: The first part is called 'the main study' and the second part is called 'the extension study'. In the main study participants will either get CagriSema (a study medicine) or placebo (a dummy medicine that looks like CagriSema but has no active ingredient). Which treatment participants get is decided by chance. Participants are two times more likely to get CagriSema than placebo. If participants get CagriSema in the main study, participants will continue on CagriSema in the extension study. Which dose of CagriSema participants will continue on is decided by chance. If participants get placebo in the main study, participants will get CagriSema in the extension study. Participants will take one injection of study medicine once a week. The study will last for about 3 years and 3 months.

ELIGIBILITY:
key Inclusion Criteria:

* Male or female (sex at birth).
* Age 18 years or above at the time of signing the informed consent.
* BMI ≥ 30.0 kilogram per square meter (kg/m^2) at screening.
* Participant has a wish to lose at least 25% of body weight within 80 weeks from randomisation.

key Exclusion Criteria:

* Glycated haemoglobin (HbA1c) ≥ 6.5% (48 millimole per mole [mmol/mol]) as measured by the central laboratory at screening.
* History of type 1 or type 2 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-10-17 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to week 80
  Measured as percentage change.

SECONDARY OUTCOMES:
Number of participants who achieve greater than or equals (≥) 20% weight reduction | From baseline (week 0) to week 80
  Measured as count of participants.
Number of participants who achieve ≥ 25% weight reduction | From baseline (week 0) to week 80
  Measured as count of participants.
Number of participants who achieve ≥ 30% weight reduction | From baseline (week 0) to week 80
  Measured as count of participants.
Number of participants who achieve normal body mass index (BMI) (18.5 kilograms per meter square (kg/m^2) less than or equal to (≤ ) BMI < 25 kg/m^2) | From baseline (week 0) to week 80
  Measured as count of participants.
Number of participants who achieve BMI < 30 kg/m^2 | From baseline (week 0) to week 80
  Measured as count of participants.
Change in waist circumference | From baseline (week 0) to week 80
  Measured as centimeter (cm).
Change in systolic blood pressure | From baseline (week 0) to week 80
  Measured as millimeters of mercury (mmHg).
Ratio to baseline in C-reactive protein (CRP) | From baseline (week 0) to week 80
  Measured as ratio.
Ratio to baseline in lipids: non-high density lipoprotein (HDL) cholesterol | From baseline (week 0) to week 80
  Measured as ratio.
Ratio to baseline in lipids: triglycerides | From baseline (week 0) to week 80
  Measured as ratio.
Ratio to baseline in lipids: HDL | From baseline (week 0) to week 80
  Measured as ratio.
Change in impact of weight on quality of life-lite for clinical trials (IWQOL-Lite-CT) physical function score | From baseline (week 0) to week 80
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Physical function score ranges from 0 to 100, with higher scores indicating better levels of functioning.
Change in short form (SF)-36v2 physical function | From baseline (week 0) to week 80
  Measured as score on a scale. The SF-36v2 acute measures health-related quality of life (HRQOL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 acute scores are norm-based scores, i.e. transformed to a scale where the 2009 United States general population has a mean of 50 and a standard deviation of 10. Physical functioning score ranges from 19.0-57.6, with higher scores indicating better functional health and well-being.
Change in IWQOL-Lite-CT physical function for subgroup with poor physical functioning at baseline (according to patient global impression of status [PGI-S]) | From baseline (week 0) to week 80
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Physical function score ranges from 0 to 100, with higher scores indicating better levels of functioning. PGI-S at baseline is used to define the subgroup with "poor" physical function in IWQOL-Lite-CT.
Change in SF-36v2 physical function for subgroup with poor physical functioning at baseline (according to PGI-S) | From baseline (week 0) to week 80
  Measured as score on a scale. SF-36v2 acute measures HRQOL. The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 acute scores are norm-based scores, i.e. transformed to a scale where the 2009 United States general population has a mean of 50 and a standard deviation of 10. Physical functioning score ranges from 19.0-57.6, with higher scores indicating better functional health and well-being. PGI-S at baseline is used to define the subgroup with "poor" physical function in SF-36V2.
Number of participants who achieve ≥ 5% weight reduction | From baseline (week 0) to week 80
  Measured as count of participants.
Number of participants who achieve ≥ 10% weight reduction | From baseline (week 0) to week 80
  Measured as count of participants.
Number of participants who achieve ≥ 15% weight reduction | From baseline (week 0) to week 80
  Measured as count of participants.
Change in waist to height ratio | From baseline (week 0) to week 80
  Measured as ratio.
Change in waist to hip ratio | From baseline (week 0) to week 80
  Measured as ratio.
Number of participants with reduction in weight category | From baseline (week 0) to week 80
  Measured as count of participants. Reduction in weight categories: underweight, BMI < 18.5 kg/m^2; normal weight 18.5 kg/m^2 ≤ BMI < 25 kg/m^2; overweight 25 kg/m^2 ≤ BMI < 30 kg/m^2; obesity class I 30 kg/m^2 ≤ BMI < 35 kg/m^2; obesity class II 35 kg/m^2 ≤ BMI < 40 kg/m^2; obesity class III BMI ≥ 40 kg/m^2.
Change in diastolic blood pressure | From baseline (week 0) to week 80
  Measured as mmHg.
Ratio to baseline in lipids: total cholesterol | From baseline (week 0) to week 80
  Measured as ratio.
Ratio to baseline in lipids: low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to week 80
  Measured as ratio.
Ratio to baseline in lipids: very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to week 80
  Measured as ratio.
Ratio to baseline in lipids: free fatty acids | From baseline (week 0) to week 80
  Measured as ratio.
Change in control of eating questionnaire (CoEQ): craving control score | From baseline (week 0) to week 80
  Measured as score on a scale. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving control subscale, the subscale score is reversed so that a higher score represents a greater level of craving control.
Change in CoEQ: positive mood score | From baseline (week 0) to week 80
  Measured as score on a scale. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the Positive Mood subscale, item 6 'How anxious have you felt?' is reversed.
Change in CoEQ: craving for sweets score | From baseline (week 0) to week 80
  Measured as score on a scale. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving sweets food subscale, higher score represents a greater level of craving.
Change in CoEQ: craving for savoury score | From baseline (week 0) to week 80
  Measured as score on a scale. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving savoury food subscale, higher score represents a greater level of craving.
Change in CoEQ: hunger score | From baseline (week 0) to week 80
  Measured as score on a scale. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the hunger subscale, higher score represents a greater level of craving.
Change in CoEQ: satiety score | From baseline (week 0) to week 80
  Measured as score points. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the satiety subscale, higher score represents a greater level of craving.
Change in IWQOL-Lite-CT: physical score | From baseline (week 0) to week 80
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Physical score ranges from 0 to 100, with higher scores indicating better levels of functioning.
Change in IWQOL-Lite-CT: psychosocial score | From baseline (week 0) to week 80
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Psychosocial score ranges from 0 to 100, with higher scores indicating better levels of functioning.
Change in IWQOL-Lite-CT: total score | From baseline (week 0) to week 80
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Total score ranges from 0 to 100, with higher scores indicating better levels of functioning.
Change in SF-36v2 health survey acute: physical component summary score | From baseline (week 0) to week 80
  Measured as score on a scale. The SF-36v2 acute measures HRQOL. The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 acute scores are norm-based scores, i.e. transformed to a scale where the 2009 United States general population has a mean of 50 and a standard deviation of 10. The physical component summary score ranges from 6.1-79.7, with higher scores indicating better functional health and well-being.
Change in SF-36v2 health survey acute: mental component summary | From baseline (week 0) to week 80
  Measured as score on a scale. The SF-36v2 acute measures HRQOL. The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 acute scores are norm-based scores, i.e. transformed to a scale where the 2009 United States general population has a mean of 50 and a standard deviation of 10. The mental component summary score ranges from -3.8-78.7, with higher scores indicating better functional health and well-being.
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to week 80
  Measured as count of events.
Number of treatment emergent serious adverse events (TESAEs) | From baseline (week 0) to week 80
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (46):
- United States (46):
  - FDRC, Costa Mesa, California
  - Linda Vista Health Care Ctr, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Northeast Research Institute, Fleming Island, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - South Broward Research LLC, Miramar, Florida
  - Florida Inst For Clin Res LLC, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Cnt for Diab,Obes, and Metab, Pembroke Pines, Florida
  - Hope Clin Res & Wellness, Conyers, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Endeavor Health, Skokie, Illinois
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Amicis Centers of Clinical Research, St Louis, Missouri
  - Mercury Str Med Grp, PLLC, Butte, Montana
  - Southgate Medical Group, LLP, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Medication Mgmnt, LLC_Grnsboro, Greensboro, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare_NC, Raleigh, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - New Venture Medical Research, Wadsworth, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - Coastal Carolina Res Ctr, North Charleston, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Amarillo Medical Specialists, Amarillo, Texas
  - Velocity Clin Res, Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Radiance Clinical Research, Lampasas, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Northeast Clinical Research of San Antonio, Schertz, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Health Res of Hampton Roads, Newport News, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Rainier Clin Res Ctr Inc, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com